CLINICAL TRIAL: NCT02385604
Title: CT-PET for Prediction of Histopathologic Response, Nodal Status and Oncologic Outcome Following Neoadjuvant Chemoradiation for Esophageal Cancer
Brief Title: The Predictive Value of CT-PET in Esophageal Cancer
Status: Completed | Type: Observational
Sponsor: St. James's Hospital, Ireland (Other)
Responsible Party: Principal Investigator, Dr Jessie A Elliott, Surgical Research Fellow, St. James's Hospital, Ireland
Other Study IDs: 12/009/2011
Record Dates: First submitted 2015-03-02; First posted 2015-03-11 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-03

CONDITIONS: Esophageal Neoplasms
Keywords: Positron-Emission Tomography; Neoadjuvant Therapy; Chemoradiotherapy; Esophagectomy; Response Evaluation Criteria in Solid Tumors; Treatment Outcome; Survival; Recurrence; Disease-Free Survival; Progression-Free Survival; Prognosis; Neoplasm Grading; Adenocarcinoma; Squamous Cell Carcinoma; Neoplasm Metastasis
MeSH Terms: conditions — Esophageal Neoplasms; Recurrence; Adenocarcinoma; Carcinoma, Squamous Cell; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A major focus of research in oncology is to identify patients who, following induction therapy, have a complete pathologic response, presenting opportunities for novel trials, including extended therapy or non-operative approaches, in addition to identifying cohorts who are resistant to the neoadjuvant therapy. The current gold standard for determining response to CRT is pathological evaluation following surgical resection, in particular the Mandard Tumour Regression Grade (TRG) or some modification thereof. At this time, however, there is no preclinical early response or post-treatment biomarker, nor endoscopic or radiologic assessment that predicts pathologic response prior to surgical resection.The aim of this study is to determine the accuracy of CT-PET for prediction of histopathologic response and/or oncologic outcome for patients with esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced esophageal or junctional neoplasm
* Histologically confirmed adenocarcinoma or squamous cell carcinoma
* Scheduled to undergo nCRT followed by surgery as per multidisciplinary Tumor Board
* CT-PET at diagnosis of malignancy (within 2 weeks from diagnosis), performed at study Center
* CT-PET 4-6 weeks after completion of nCRT, prior to surgical resection

Exclusion Criteria:

* Incomplete data, patient lost to follow-up
* Scans performed at alternate Center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Records for all patients with locally advanced esophageal and junctional tumors undergoing potentially curative multimodal therapy between November 2008 and November 2014 will be assessed.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | Undetermined
Disease-free survival | Undetermined

SECONDARY OUTCOMES:
Histopathologic response | Undetermined
  Mandard tumor regression grade, ypT, ypN stage

CONTACTS AND LOCATIONS:
Overall Officials: John V Reynolds, MCh FRCS, Principal Investigator — Department of Surgery, St. James's Hospital
Locations (1):
- Department of Surgery, St. James's Hospital, Dublin, Ireland

REFERENCES:
- [Background] Donohoe CL, O'Farrell NJ, Grant T, King S, Clarke L, Muldoon C, Reynolds JV. Classification of pathologic response to neoadjuvant therapy in esophageal and junctional cancer: assessment of existing measures and proposal of a novel 3-point standard. Ann Surg. 2013 Nov;258(5):784-92; discussion 792. doi: 10.1097/SLA.0b013e3182a66588. PMID 24045450
- [Background] Piessen G, Petyt G, Duhamel A, Mirabel X, Huglo D, Mariette C. Ineffectiveness of (1)(8)F-fluorodeoxyglucose positron emission tomography in the evaluation of tumor response after completion of neoadjuvant chemoradiation in esophageal cancer. Ann Surg. 2013 Jul;258(1):66-76. doi: 10.1097/SLA.0b013e31828676c4. PMID 23470576
- [Result] Elliott JA, O'Farrell NJ, King S, Halpenny D, Malik V, Muldoon C, Johnston C, Reynolds JV. Value of CT-PET after neoadjuvant chemoradiation in the prediction of histological tumour regression, nodal status and survival in oesophageal adenocarcinoma. Br J Surg. 2014 Dec;101(13):1702-11. doi: 10.1002/bjs.9670. Epub 2014 Oct 28. PMID 25351460